CLINICAL TRIAL: NCT00713661
Title: Non-randomised, Open, Multi-center Trial Evaluating Feasibility and Safety of TachoSil® Application on a Colorectal Anastomosis.
Brief Title: Evaluation of TachoSil® Application on a Colorectal Anastomosis (TC-029-IM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nycomed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TC-029-IM; 2007-007254-62 (EudraCT Number)
Record Dates: First submitted 2008-07-07; First posted 2008-07-11 (Estimated); Results first posted 2012-03-02 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-02

CONDITIONS: Colorectal Anastomosis
Keywords: Colorectal Anastomosis; Colorectal Resection; Tachosil
MeSH Terms: interventions — TachoSil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TachoSil® (Experimental)
  Interventions: Drug: TachoSil®

INTERVENTIONS:
Drug: TachoSil® — Sterile, ready-to-use, absorbable sponge for intra-operative topical application. It consists of an equine collagen sponge coated with the fibrin glue components human fibrinogen and human thrombin.
  Surgery was performed according to the hospitals' local standards. When the anastomosis was performed, all enrolled subjects had TachoSil® applied around the anastomotic line. TachoSil® was therefore an add-on therapy.

SUMMARY:
The primary objective is to evaluate if the application of TachoSil® on a colorectal anastomosis is feasible and safe.

The secondary objective is to establish and describe optimal application methods to be used for educational purposes in future trials.

ELIGIBILITY:
Inclusion Criteria - at screening:

* Has the patient given informed consent according to local requirements before any trial-related activities? A trial-related activity is any procedure that would not have been performed during the routine management of the subject.
* Is the subject 18 years of age or above?
* Is the subject scheduled for elective resection of the rectum?
* Is a colorectal anastomosis below the peritoneal reflexion planned?

For females of childbearing potential:

* Does the patient use an acceptable contraceptive method (contraceptive pills, injection of prolonged gestagen, subdermal implantation, hormonal vaginal devices, transdermal patches or intrauterine device (IUD))?
* Is the blood or urine pregnancy test negative?

Exclusion Criteria -at screening:

* Is the subject scheduled for emergency resection of the rectum?
* Does the subject suffer from inflammatory bowel diseases?
* Does the subject have a history of hypersensitivity reactions after application of human fibrinogen, human thrombin and/or collagen of any origin?
* Has the subject participated in any other trial with an investigational medical product (IMP) or device within 30 days before inclusion in this trial?
* Does the subject participate or plan to participate in another clinical trial during the trial period?

For females of childbearing potential:

• Is the subject pregnant or breast feeding?

Exclusion - peroperative

* Was an anastomosis performed differently from what was defined in the inclusion criteria?
* Did the subject receive any fibrin sealant/glue, excluding TachoSil® , during surgery?

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nycomed Clinical Trial Operations, Study Chair — Headquarters
Locations (3):
- Investigational site, Berlin, Germany
- Investigational site, Utrecht, Netherlands
- Investigational site, Dartford, Kent, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were divided into
  * Surgery method: open or laparoscopic
  * Location of the anastomosis:
    * anastomotic line in the low segment (approx. 0-5 cm from the anal verge)
    * anastomotic line in the mid or upper segment (approx. 5-12 cm from the anal verge)
Groups:
- Group 1: Open Surgery Lower: Open colorectal resection. The anastomotic line in the low segment approximately 0-5 cm from the anal verge.
- Group 2: Open Surgery Middle/Upper: Open colorectal resection. The anastomotic line in the middle/upper segment 5-12 cm from the anal verge.
- Group 3: Laparoscopic Surgery Lower: Laparoscopic colorectal resection. The anastomotic line in the low segment approximately 0-5 cm from the anal verge.
- Group 4: Laparoscopic Surgery Middle/Upper: Laparasocopic colorectal resection. The anastomotic line in the mid/upper segment 5-12 cm from the anal verge.
Period: Overall Study
Arm/Group | Group 1: Open Surgery Lower | Group 2: Open Surgery Middle/Upper | Group 3: Laparoscopic Surgery Lower | Group 4: Laparoscopic Surgery Middle/Upper
Started | 7 | 9 | 4 | 5
Completed | 7 | 9 | 4 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Open Surgery Lower | Group 2: Open Surgery Middle/Upper | Group 3: Laparoscopic Surgery Lower | Group 4: Laparoscopic Surgery Middle/Upper | Total
Number analyzed (Participants) | 7 | 9 | 4 | 5 | 25
Age Continuous [Mean (Standard Deviation); unit: years] | 63.7 (8.5) | 64.6 (12.8) | 68.5 (9.9) | 65.2 (12.0) | 65.1 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 0 | 5 | 8
  Male | 7 | 6 | 4 | 0 | 17

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint is the Feasibility of the TachoSil® Application, Reported by the Combined Assessment of the Investigator and External Assessor
Description: Evaluation of feasibility was assessed by investigator after application of the TachoSil® sponge on the anastomosis. A feasible application implied that the entire TachoSil® adhered and covered at least 1cm beyond the margins of the anastomotic line and that if more than one sponge was used, they overlapped by at least 1 cm. The score was assisted by video recording. To ensure an independent assessment, the recording was assessed by an external, blinded assessor. In case of discrepancies between the assessment of the investigator and the assessor, the application was regarded as not feasible.
Time Frame: Day of surgery
Population: ITT + Safety Analysis Set.
  All applications recorded as "not feasible" by external assessor was because he was not able to see it all the way around the anastomosis. The implication is that the primary endpoint was not really reporting the true feasibility, as it was hindered due to technical/practical problems recording the whole anastomosis.
Measure: Number; unit: participants
Arm/Group | Group 1: Open Surgery Lower | Group 2: Open Surgery Middle/Upper | Group 3: Laparoscopic Surgery Lower | Group 4: Laparoscopic Surgery Middle/Upper
Number analyzed (Participants) | 7 | 9 | 4 | 5
participants
  Video not available | 1 | 2 | 1 | 2
  Feasible | 2 | 5 | 2 | 3
  Not feasible | 4 | 2 | 1 | 0

2. Secondary Outcome: The Secondary Endpoint is the Feasibility of the TachoSil® Application, Assessed by the Investigator.
Description: Evaluation of feasibility was assessed by investigator after application of the TachoSil® sponge on the anastomosis. A feasible application implied that the entire TachoSil® adhered and covered at least 1cm beyond the margins of the anastomotic line and that if more than one sponge was used, they overlapped by at least 1 cm. The score was assisted by video recording.
Time Frame: Day of surgery
Population: Data are presented for the 25 subjects treated with TachoSil®. They constitute the intention-to-treat (ITT) and the safety analysis set.
Measure: Number; unit: participants
Arm/Group | Group 1: Open Surgery Lower | Group 2: Open Surgery Middle/Upper | Group 3: Laparoscopic Surgery Lower | Group 4: Laparoscopic Surgery Middle/Upper
Number analyzed (Participants) | 7 | 9 | 4 | 5
participants
  Feasible | 6 | 9 | 4 | 5
  Not feasible | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The safety population consists of all 25 subjects that received trial treatment.
  SAE/AE assessment by neutral questioning "Have you experienced any health problems since the last contact?" by the investigator at each contact (visit or phone).
Arm/Group | Group 1: Open Surgery Lower | Group 2: Open Surgery Middle/Upper | Group 3: Laparoscopic Surgery Lower | Group 4: Laparoscopic Surgery Middle/Upper
Serious Adverse Events (participants affected / at risk) | 3/7 | 1/9 | 3/4 | 0/5
Other Adverse Events (participants affected / at risk) | 3/7 | 3/9 | 1/4 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Open Surgery Lower (N=7) | Group 2: Open Surgery Middle/Upper (N=9) | Group 3: Laparoscopic Surgery Lower (N=4) | Group 4: Laparoscopic Surgery Middle/Upper (N=5)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — SAE was reported as not related to TachoSil®.
Small bowel obstruction caused by adhesions requiring small bowel resection done open (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — SAE was reported as not related to TachoSil®.
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — SAE was reported as not related to TachoSil®.
Anastomotic leakage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — SAE was reported as not related to TachoSil®.
Minor anastomotic leakage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — SAE was reported as not related to TachoSil®.
Stomaprolaps (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — SAE was reported as not related to TachoSil®.
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — SAE was reported as not related to TachoSil®.
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — SAE was reported as not related to TachoSil®.
Pelvic haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — SAE was reported as not related to TachoSil®.
Presacral haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — SAE was reported as not related to TachoSil®.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Open Surgery Lower (N=7) | Group 2: Open Surgery Middle/Upper (N=9) | Group 3: Laparoscopic Surgery Lower (N=4) | Group 4: Laparoscopic Surgery Middle/Upper (N=5)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After publication of the results or 24 months after Clinical Trial Report has been finalised, whichever comes first, Nycomed acknowledge the Investigator's rights to publish results from this trial. Any such scientific paper, presentation, communication, or other information concerning the investigation described in this protocol, must be submitted to Nycomed prior to submission for publication/presentation for review. Review comments will be given within a month from receipt of the manuscript.